CLINICAL TRIAL: NCT05499741
Title: Piloting Forehead Temperature-Regulating Therapy for Insomnia in Adults With Tourette's Disorder
Brief Title: Forehead Temperature-Regulating Therapy for Insomnia in Adults With Tourette's Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Emily J. Ricketts, PhD, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-000432; 30464 (Other Grant/Funding Number: Brain and Behavior Research Foundation)
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Tourette's Disorder; Insomnia
Keywords: tics; insomnia; sleep; temperature; device
MeSH Terms: conditions — Tourette Syndrome; Sleep Initiation and Maintenance Disorders; Tics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Forehead Temperature-Regulating Therapy (Experimental): Forehead Temperature-Regulating Therapy
  Interventions: Device: Forehead Temperature-Regulating Therapy

INTERVENTIONS:
Device: Forehead Temperature-Regulating Therapy — A forehead thermal therapy device will be used nightly for the duration of each sleep period for four weeks. This device includes a bedside unit and a pump to transport thermal fluid to a bladder, affixed to the forehead with a headband. The bladder circulates fluid over the forehead at adjustable temperatures ranging from 57-61 °F.
  Other Names: Ebb CoolDrift Versa

SUMMARY:
The primary aim of the present research project is to investigate the preliminary effects of four weeks of forehead temperature-regulating therapy on insomnia in adults with Tourette's disorder and co-occurring insomnia disorder. This project will also examine the effects of the device on depression, anxiety, and daytime sleepiness, and explore its effects on tic severity.

DETAILED DESCRIPTION:
Tourette's disorder is a neurological condition marked by multiple motor tics and one or more vocal tics present for longer than one year, and neural dysfunction within the frontal region of the brain. Sleep disturbance, particularly insomnia, is common in Tourette's disorder. Existing treatments (medication, behavior therapy) for Tourette's disorder do not benefit everyone. The sleep-wake cycle, which may overlap with Tourette's disorder with respect to underlying brain-based deficits, provides a key target for tailored intervention. Forehead temperature-regulating therapy, designed to treat insomnia through targeting underlying brain-based functioning, provides one such intervention. Therefore, the aim of the present investigation is to examine the preliminary effects of forehead temperature-regulating therapy on 1) insomnia, 2) depression, anxiety and daytime sleepiness, and 3) tic severity in adults with Tourette's disorder and co-occurring insomnia disorder.

Participation involves an initial assessment, during which an evaluator will screen for psychiatric and sleep disorder diagnosis, tic severity, and cognitive functioning. Participants will rate sleep apnea risk, insomnia severity, depression, anxiety, and daytime sleepiness. Participants will then monitor sleep for seven consecutive nights by wearing a wrist actigraph (sleep watch) and completing a sleep diary. Participants will then complete a pre-treatment evaluation, during which an evaluator will reassess tic severity, and participants will rate depression, anxiety, and daytime sleepiness. After the pre-treatment evaluation, participants will use a forehead temperature-regulating therapy device nightly for four weeks. Participants will use the actigraph and sleep diary to monitor sleep continuously for the remainder of the study. Following the intervention, participants will complete a post-treatment assessment involving clinician-rated tic severity interview, and re-rating of depression, anxiety, and daytime sleepiness measures. Findings will help researchers determine the degree to which non-medication treatments are helpful for insomnia in people with Tourette's disorder.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of Tourette's disorder
* DSM-5 diagnosis of Insomnia disorder
* Yale Global Tic Severity Scale Score ≥ 14 for Tourette's disorder or ≥ 10 for persistent motor tic disorder or persistent vocal tic disorder
* Insomnia Severity Index score > 14
* Sleep efficiency ≤ 85 per cent on 50 percent or greater nights over monitoring week, per Consensus Sleep Diary
* Age of 18 to 50 years
* English fluency

Exclusion Criteria:

* Current or lifetime diagnosis of bipolar disorder, psychosis, or pervasive developmental disorder
* Suicidality, severe depression or anxiety, or alcohol or substance dependence present within the past 6 months
* Moderate to severe sleep apnea risk per score of ≥ 3 on the Stop-Bang Questionnaire
* current diagnosis of Narcolepsy
* Wechsler Abbreviated Scale for Intelligence-Second Edition IQ score < 80
* Changes in prescribed or over-the-counter medications for sleep within prior month and planned during the study
* Changes in tic or other psychotropic medication within prior month and planned during study
* Caffeine use > 3 cups per day
* Behavior therapy for tics or sleep within prior 3 months
* Travel across > 2 time zones in prior month
* Shift work, or irregular sleep schedule (i.e., nightly variation of > 3 hours in bedtime or wake time, or time in bed duration < 5.5 or > 10 hours per night)
* Raynaud's disease or severe cold sensitivity
* Other major medical or neurological condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Actigraphy - Sleep Onset Latency | 5 weeks
  Sleep onset latency will be measured via a wrist actigraph and is defined as duration in minutes between time in bed and sleep onset. An actigraph (Actiwatch Spectrum PRO, Philips Respironics, Amsterdam, Netherlands), worn on the non-dominant wrist, will record daily and nightly movement/activity. Actigraphs will be set to record movements in 30-second epochs. Actigraphy data will be converted into sleep-wake scores guided by sleep diary bed times and rise times.
Actigraphy - Wake After Sleep Onset | 5 weeks
  Wake after sleep onset will be measured via a wrist actigraph and is defined as the total number of minutes spent awake following sleep onset. An actigraph (Actiwatch Spectrum PRO, Philips Respironics, Amsterdam, Netherlands), worn on the non-dominant wrist, will record daily and nightly movement/activity. Actigraphs will be set to record movements in 30-second epochs. Actigraphy data will be converted into sleep-wake scores guided by sleep diary bed times and rise times.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale (DASS)-21 - Depression | 5 weeks
  The DASS-21 (Lovibond & Lovibond, 1995) is a 21-item self-report measure of depression, anxiety, and stress symptoms in the past week. Items are rated according to a 0- to- 3 scale and summed to yield independent depression, anxiety, and stress scores. Subscale scores are normed by multiplying them by two. Higher scores indicate increased negative affect.
Depression Anxiety Stress Scale (DASS)-21 - Anxiety | 5 weeks
  The DASS-21 (Lovibond & Lovibond, 1995) is a 21-item self-report measure of depression, anxiety, and stress symptoms in the past week. Items are rated according to a 0- to- 3 scale and summed to yield independent depression, anxiety, and stress scores. Subscale scores are normed by multiplying them by two. Higher scores indicate increased negative affect.
Epworth Sleepiness Scale (ESS) | 5 weeks
  The ESS (Johns, 1991) is an 8-item self-reported measure of daytime sleepiness assessing potential for dozing or falling asleep across 8 situations. Items are rated on a 0- to- 3-scale and summed to yield a total score ranging from 0 to 24. Higher scores indicated increased daytime sleepiness.

OTHER OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) - Total Tic Severity Score | 5 weeks
  The YGTSS (Leckman et al., 1989) is a clinician-rated measure of tic symptom severity and tic-related impairment. Tic severity is assessed across number, frequency, intensity, complexity, and interference. Ratings are summed to produce separate scores for motor tics (0-25) and vocal tics (0-25), which are then summed to produce a total tic severity score (0-50).

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Ricketts, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Semel Institute for Neuroscience and Human Behavior, University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888